CLINICAL TRIAL: NCT05911009
Title: A Prospective, Double-blind, Randomized, Parallel Group, Placebo Controlled, Multicentre, Phase II Study to Investigate the Efficacy, GPCR Autoantibody Neutralizing Effect, Safety, and Tolerability of BC 007 in Participants With Long COVID
Brief Title: To Investigate Efficacy, Pharmacodynamics, and Safety of BC 007 in Participants With Long COVID
Acronym: BLOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Berlin Cures GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBC007C401; 2022-003452-14 (EudraCT Number)
Record Dates: First submitted 2023-06-15; First posted 2023-06-20 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Long Covid
Keywords: Long Covid; Autoantibodies; Post-acute COVID-19 syndrome; BC 007; PASC
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, parallel group, placebo controlled, multicentric
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1350mg BC 007 solution for infusion for 75-minutes intravenous infusion (Experimental)
  Interventions: Drug: BC 007 or matching placebo
- 0.9% NaCl solution for infusion for 75-minutes intravenous infusion (Placebo Comparator)
  Interventions: Drug: BC 007 or matching placebo
- 1900mg BC 007 solution for infusion for 105-minutes intravenous infusion (Experimental)
  Interventions: Drug: BC 007 or matching placebo
- 0.9% NaCl solution for infusion for 105-minutes intravenous infusion (Placebo Comparator)
  Interventions: Drug: BC 007 or matching placebo

INTERVENTIONS:
Drug: BC 007 or matching placebo — Participants will be treated with two infusions of BC 007 or placebo two weeks apart, according to a double-blind design

SUMMARY:
This study is an interventional, randomized, multinational, multicenter, double-blind, phase 2 study with a follow-up period of 90 days.

The intension of this clinical trial is to investigate the long-term sequelae (named Long COVID syndrome; post COVID or PASC) of an infection with Corona Virus Type 2 that has resulted in a condition known as Severe Acute Respiratory Syndrome Corona Virus Type 2 (SARS-CoV-2).

The purpose of this study is to evaluate the efficacy and safety of BC 007 as a treatment for long-lasting COVID-symptoms in patients who were neither intubated nor supported with extracorporeal blood oxygenation (ECMO) during their acute COVID-19 infection.

The study drug acts by neutralizing functional autoantibodies directed against G-protein coupled receptors (GPCRs).

Neutralization of the autoantibodies is expected to induce a beneficial effect on symptoms typically seen in patients with long COVID syndrome.

Functional autoantibodies are proteins belonging to the class of G-type immunoglobulins that can be synthesized by activation of the immune system and can induce various pathogenic activities by binding to one of the extracellular loops of G-proteins (GPCR-AAB).

The study consists of a screening phase of up to 35 days, treatment (two administrations by intravenous infusion at two-week intervals either with the study drug (BC 007) or with placebo (NaCl 0.9%), with an initial follow-up period of 15 days after each administration and an extended follow-up period of 60 days.

Patients are required to visit the study center for follow-up visits at specified intervals.

For the entire study duration of 125 days from screening to the end of the study, 8 site visits are planned.

ELIGIBILITY:
Inclusion Criteria:

Participant is eligible to be included in the study only if all the following criteria apply:

1. The participant provides written informed consent prior to any clinical study-specific procedures.
2. The participant is a male or female, ≥18 years of age, at the time of signing the informed consent form.
3. All male and female participants of childbearing potential must be willing to use effective methods of contraception from the start of Screening until EOS (Day 90). Male participants must refrain from donating sperm during this period.
4. Acute phase of COVID-19 ended at least 3 months prior to dosing.
5. The participant has a confirmed negative SARS-CoV-2 test result (polymerase chain reaction [PCR] test) at screening.
6. The participant provides a documented positive SARS-CoV-2 test result (reverse transcriptase [RT]-PCR or rapid antigen test) at Screening. For participants with long COVID symptoms who cannot provide certified evidence, a positive antibody test for nucleocapsid protein IgG must demonstrate a history of SARS CoV 2 infection; this test can be performed as part of the Screening procedure. The participant reports persistence or new onset of symptoms after a SARS-CoV-2 infection, with these symptoms lasting for at least 2 consecutive months (being persistent, recurrent, or of varying severity within that period) with no other explanation, as defined by WHO, and not being present prior to COVID-19 infection.
7. Participant is screened positive for GPCR-AAB activity by Berlin Cures laboratory.
8. Participant has not been intubated or received ECMO support during their acute COVID-19 infection.
9. Participant screens positive for fatigue (FACIT-FS score <35) and presents with at least one additional symptom from the symptom score sheet (COA) which has persisted for more than 12 weeks.
10. Participant is not on any permanent medication(s) to treat chronic diseases that existed prior to COVID 19 infection. Exceptions are clinically stable conditions, which do not affect the study assessments and may be allowed as judged by the Investigator after discussion with the medical monitor. Clinically unstable is defined as a diagnosis or condition requiring changes in disease management within 2 months prior to start of Screening and includes ongoing workup of an undiagnosed illness that could lead to a new diagnosis or condition. Concomitant treatment may be permitted, if

    * A treatment (type and dose) remained unchanged within the 2 months before the start of Screening.
    * No change in treatment is expected or required between Screening visit and Day 30 of the study.
    * A treatment does not affect any of the study assessments, in particular by (e.g.,) causing fatigue or by impairing concentration ability.

    As judged by the Investigator and after discussion with the medical monitor, possible allowed concomitant medications include but are not limited to:
    * Antihypertensives (β-blockers are NOT allowed)
    * Lipid lowering agents.
    * Antidiabetics (insulin is NOT allowed)
    * Thyroid hormone replacement.
    * Topical treatments.
    * Low dose acetylsalicylic acid (up to 100 mg/day).
    * Ivabradine.
11. Participant reports that his/her activity level was not impaired prior to acute COVID-19 infection.

Exclusion Criteria:

Participant is excluded from the study if any of the following criteria apply:

1. Postural Orthostatic Tachycardia Syndrome existing prior to the initial SARS CoV 2 infection leading to long COVID, as per medical history. History or evidence of any clinically significant cardiovascular disease.
2. Any history or presence of gastrointestinal, endocrinologic (Type 1 diabetes,), cardiovascular, haematologic, hepatic, immunologic, metabolic (specifically gout), urologic, pulmonary (asthma), neurologic, dermatologic, renal and/or other major disease , as judged by the Investigator before SARS-CoV-2 infection. Other clinically stable conditions, which do not affect the study assessments may be allowed as judged by the Investigator after discussion with the medical monitor.

   Possible allowed diseases are (if stable and well-controlled) include but are not limited to:
   * Respiratory disorders (e.g., asthma-like) that first appear with long COVID.
   * Mild hypertension (<160 mmHg systolic, <100 mmHg diastolic) without known organ or vessel damage.
   * Non-insulin-dependent diabetes mellitus without known organ or vessel damage.
   * Glaucoma.
   * Hypercholesterolemia/hypertriglyceridemia.
   * Hypothyreosis
3. Participants with history of major active or chronic unstable psychiatric illness (e.g., but not limited to, depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year.
4. Any history of any other chronic neurological, or psychological disease such as, but not limited to, chronic fatigue syndrome, fibromyalgia, lupus, Sjogren's syndrome.

   Any history or presence of relevant allergic reactions (e.g., requiring hospital stay, intravenous [i.v.] treatment or treatment with systemic steroids). A participant will not be included if it is likely that seasonal allergic symptoms will require any kind of systemic treatment until Day 30 of the study.
5. Participant has a history of hypersensitivity to the study intervention or any of the excipients or to medicinal products with similar chemical structures.
6. Participant has any other condition, which in the opinion of the Investigator precludes the participant's participation in the clinical study.
7. Participant shows clinically significant abnormalities in clinical chemistry or haematology at screening, as judged by the Investigator.
8. Female participant is pregnant and/or breast feeding.
9. Participant participated in a previous clinical study (within 30 days or 5 half-lives of the investigational drug, or whichever is longer prior to start of Screening) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s),or participant previously participated in this study and received study intervention.
10. Participant is an employee of the Sponsor, or contract research organization (CRO) conducting the study.
11. Participant has a close affiliation with the investigational site, e.g., a close relative of the Investigator, dependent person (e.g., employee or student of the investigational site).
12. Participant with an estimated glomerular filtration rate <60 mL/min/1,73 m².
13. Participant has alcohol addiction or history of alcohol addiction.
14. Participant has drug addiction or history of drug addiction.
15. Any psychological, emotional problems, any disorders or resultant therapy that is likely to invalidate informed consent or limit the ability of the participant to comply with the protocol requirements.
16. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the last 5 years.
17. Participant has had comparable and prolonged symptoms after other viral infections (e.g., after Epstein-Barr virus infection, influenza, infectious mononucleosis).
18. Previous diagnosis of sleep apnoea.
19. Current use of medications with psychoactive properties that have a deleterious effect on cognition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in score on FACIT-FS scale at Day 30. | Day 30
  To compare efficacy of BC 007 (double dose 1350 mg and double dose 1900 mg) with placebo based on Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale in long COVID participants.
  FACIT-F is a five-point scale from 0 (not at all) to 4 (very much). The maximum composite scale is 52 (range 0 to 52). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
To compare GPCR AAB neutralizing effect of BC 007 1350 mg with that of placebo. | at Days 3, 15, 17, 30, 60 and Day 90 post first infusion of study intervention.
  Proportion of participants sero-converting to negative for GPCR-AAB
To compare GPCR AAB neutralizing effect of BC 007 1900 mg with that of placebo. | at Days 3, 15, 17, 30, 60 and Day 90 post first infusion of study intervention.
  Proportion of participants sero-converting to negative for GPCR-AAB
To compare GPCR-AAB neutralizing effect of BC 007 1350 mg with that of BC 007 1900 mg | at Days 3, 15, 17, 30, 60 and Day 90 post first infusion of study intervention.
  Proportion of participants sero-converting to negative for GPCR-AAB

CONTACTS AND LOCATIONS:
Overall Officials: Axel Mescheder, Dr., Study Director — CMO Berlin Cures GmbH
Locations (16):
- Austria (2):
  - Klinik Favoriten - Wiener Gesundheitsverbund, Vienna
  - Klinik Floridsdorf - Wiener Gesundheitsverbund, Vienna
- Terveystalo Helsinki Sleep Clinic, Helsinki, Nyland and Tavastehus County, Finland
- Germany (8):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Krankenhaus Havelhöhe, Berlin
- Spain (4):
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospitalario Universitario Quironsalud Madrid, Madrid
  - Hospital General de Málaga, Málaga
  - University Hospital Virgen Del Rocio S.L., Seville
- Stadtspital Zurich Waid, Zurich, Switzerland